CLINICAL TRIAL: NCT07061782
Title: Effects of Neuromuscular Reeducation Versus Post Facilitation Stretch Technique for Upper Cross Syndrome Among IT Professionals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/82
Record Dates: First submitted 2025-06-04; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): On group A hot pack 10 min on cervical area investigator will perform NEUROMUSCULAR REEDUCATION TECHNIQUE: investigator will perform this technique on tight muscles which are:
  1. levator scapulae
  2. upper trapezius
  3. pectoralis major
  4. strengthening exercises
  Interventions: Procedure: Group A
- Group B (Experimental): On group B hot pack for 10 min on cervical area investigator will perform POST FACILITATION STRETCH TECHNIQUE on tight muscles same as group A
  1. levator scapulae
  2. upper trapezius
  3. pectoralis major
  4. strengthening exercises
  Interventions: Procedure: Group B

INTERVENTIONS:
Procedure: Group A — Treatment protocol given to the both groups will be carried out for 7 sessions for 2 weeks on alternative days.
  It will consist of a 10 minute hot pack.
  Neuromuscular reeducation for following muscles. Pectoralis major Upper trapezius Levator scapulae
  Strengthening exercises of:
  Rhomboids Lower & middle trapezius Deep flexors Neuromuscular reeducation It will break adhesion result in loosen the scar tissue will increase the temperature and cause in increase of blood flow . Muscles contract when myosin pulls actin filaments together using energy from ATP shortening the muscle fiber and causing contraction. They relax when calcium is removed, allowing the filaments to slide apart muscle will return to its resting state. The continuously muscle contraction and relaxation help to loosen up and become more flexible .
  Strengthening exercises
  Arms: Group A
Procedure: Group B — Treatment protocol was given to both groups for 7 session sessions for 2 weeks on alternative days.
  It was comprises of HOT PACK for 10 minutes . Post facilitation stretch for following muscles. Pectoralis major Upper trapezius Levator scapulae
  Strengthening exercises of:
  Rhomboids Lower & middle trapezius Deep flexors
  Post facilitation stretch :
  Post Facilitation Stretch is an isometric Contraction in which he participants were instructed to contract the muscles to the maximum voluntary capacity that involves first putting the target muscle through a high-intensity isometric contraction (roughly 75-100% of maximal effort) for 5-10 seconds, and then quickly and continuously passively stretching the same muscle for at least 10 seconds.
  Strengthening exercises
  Arms: Group B

SUMMARY:
This study is a randomised control trial and the purpose of this study is to determine the "Effects of Neuromuscular Reeducation Versus Post Facilitation Stretch Technique for Upper Cross Syndrome among IT professionals

DETAILED DESCRIPTION:
The purpose of this study is to determine the "Effects of Neuromuscular Reeducation Versus Post Facilitation Stretch Technique for Upper Cross Syndrome among IT professionals

Investigator will make 2 groups control and treatment group . investigator will give NMR technique to treatment group and PFS technique to control group in patients with upper cross syndrome.

first investigator will take base line readings of cervical ROM by using goniometer , NPRS AND neck diasbilty index.

after 2 weeks of treatment again investigator will take same readings and compare both readings.

with techniques investigator will also perform strengthning excercise of weal muscles for both groups

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

IT profressionals 20 - 40 years Both genders Diagnosed UCS Pain from 2 months Minimum 4 - 6 hours working

Exclusion Criteria:

* History of cervical spine Fracture Trauma to neck

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Upper cross syndrome pain | baseline and after 2 weeks
  Assessed using the Numeric Pain Rating Scale (NPRS). Patient is asked to rate the intensity of pain in numbers ranging from 0 to 10. This self-assessment tool uses an 11 point numeric scale ranging from 0 (no pain ) to 10 (worst pain)
Posture and Muscle Balance | baseline and after 2 weeks
  Assessed using the Neck disability index (NDI) It is a self- rating questionnaire includes ten items . Each item in the neck disability index has six different options or scores indicating the progressive levels of pain or activity of daily life limitations. Item are scored from 0 to 5 where 0 indicates no pain or limitation and 5 indicates maximum possible pain and limitation. Investigator use Janda approach to check the muscles tightness and weaknesss For tight muscles investigator use Muscle length test For weak muscles investigator use Muscle strength test
Cervical range of motion | baseline and after 2 weeks
  Flexion, extension, lateral flexion, and rotation measured using a goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan